CLINICAL TRIAL: NCT06770023
Title: A Pilot Study of Transseptal ECMO With the Protek Solo Cannula in Lung Transplant Candidates With Right Heart Failure From Pulmonary Hypertension
Brief Title: Bridge to Lung Transplant With Trans-septal Extra-corporeal Membrane Oxygenation (ECMO) for Right Heart Failure From Pulmonary Hypertension
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ian Makey, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-000660
Record Dates: First submitted 2025-01-06; First posted 2025-01-13 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Lung Transplant; Pulmonary Hypertension
Keywords: right heart failure, transseptal, extra-corporeal membrane oxygenation, bridge to transplant
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lung transplant patients (Experimental): Subjects will be those who are on the transplant list and progress to needing right ventricle (RV) support
  Interventions: Device: Protek Solo Transseptal Cannula

INTERVENTIONS:
Device: Protek Solo Transseptal Cannula — The Protek Solo Transseptal Cannula ECMO cannula will be placed from the right femoral vein and the drainage cannula will be placed from either the left femoral vein or the right internal jugular vein.

SUMMARY:
The purpose of this study is to determine if transseptal extra-corporeal membrane oxygenation (ECMO) can bridge pulmonary hypertension- right heart failure (PH-RVF) patients to lung transplant safely.

DETAILED DESCRIPTION:
Results will be released as a manuscript once it has gone through the peer review process. Results will be released even in the event of negative outcomes and the release will be hastened if the study is terminated early.

Medicare beneficiaries may be affected by the device under investigation if they are candidates for lung transplant. Since this is such a select group of patients, we do not expect the results of this trial to be generalizable to the general Medicare population.

ELIGIBILITY:
Inclusion Criteria

Patients that are listed for lung transplantation and have:

* PH defined as:

  * Group 1 Pulmonary arterial hypertension (PAH): Mean pulmonary artery pressure (PAP) ≥ 20 mm Hg, pulmonary capillary wedge pressure (PCWP) < 15 mm Hg, and pulmonary vascular resistance (PVR) ≥ 3 Wood units
  * Group 3 PH is defined as the presence of chronic lung disease (CLD) and/or hypoxia and mean pulmonary artery pressure (PAP) ≥ 20 mm Hg.
* Secondary PH (WHO Group 3) or diagnosis of primary PH (WHO Group 1) (to include Eisenmenger syndrome).
* Failing right ventricle function defined as:

  * a cardiac (CI) index < 2.2 L/min/m^2 despite continuous infusion of high dose inotropes defined as:
  * Inhaled nitric oxide > 20 ppm and one of the following:
  * Dobutamine > 10 ug/kg/min x 15 minutes or
  * Milrinone > 0.5 ug/kg/min x 120 minutes or
  * Epinephrine > 0.5 ug/kg/min x 15 minutes or
  * Norepinephrine > 0.5 ug/kg/min x 15 minutes and have one of the following:

    1. central venous pressure (CVP) > 15 mm Hg
    2. global RV dysfunction on echocardiography defined as one of the following:

       1. a tricuspid annular plane systolic excursion score of <14mm
       2. an RV diameter at base >42mm
       3. RV short-axis or midcavity diameter >35mm
  * Lactate greater than 3 mmol/L
  * Urine output < 0.5 ml/kg/hour
* Age > 18 years old
* BMI <35
* Informed consent signed by self or legally authorized representative.

Exclusion Criteria

* INTERMACS 1 patients (Critical cardiogenic shock patient who is "crashing and burning", has life-threatening hypotension and rapidly escalating inotropic or pressor support, with critical organ hypoperfusion often confirmed by worsening acidosis and lactate levels)
* End organ failure defined as: hepatic total bilirubin >5 mg/dL based on lab data within 24 hours prior to transseptal ECMO initiation; renal creatinine >4 mg/dLbased on lab data within the 24 hours prior to transseptal ECMO initiation
* Evidence of acute neurologic injury
* Active infection defined as two of the following WBC >12,500, positive blood culture, fever
* RA thrombus
* Thrombolysis within the previous 30 days or known existing coagulopathy such as thrombocytopenia or hemoglobin diseases such as sickle cell anemia or thalassemia
* Right heart failure from isolated pulmonary embolism
* Right heart failure from coronary artery disease or from left heart failure (WHO Type 2)
* Congenital forms of pulmonary hypertension such as tetralogy of fallot or pulmonary vein stenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Survival until transplant | 3 weeks
  Number of subjects to survive between placement of cannula and lung transplant.

SECONDARY OUTCOMES:
Number of subjects to experience adverse events | 2 months
  Adverse events are defined as: death, major bleeding, failure to achieve left atrium access, device migration and stroke.
Extra-corporeal membrane oxygenation (ECMO) support | 2 months
  Number of days after transplant on ECMO support
Dialysis | 2 months
  Number of subjects who need dialysis after transplant
Hospital Discharge | 2 months
  Number of patients that are successfully discharged from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ian Makey, MD, Principal Investigator — Mayo Clinic; Mohammad E Alomari, MD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No